CLINICAL TRIAL: NCT02196272
Title: The Efficacy of a Nurse-led Reminder Program on Therapy Adherence, Clinical Outcomes and Trust in Nurses in Diabetic Patients.
Brief Title: Nurse-led Reminder Program for Therapy Adherence, Clinical Outcomes and Trust in Nurses in Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Sanitaria Locale n. 2 - Lanciano Vasto Chieti (Other)
Responsible Party: Principal Investigator, Giancarlo Cicolini, PhD, Azienda Sanitaria Locale n. 2 - Lanciano Vasto Chieti
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAPS-001
Record Dates: First submitted 2014-07-15; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Nurse-led email program through email (Experimental): In addition to usual care and educational program, the intervention group will also receive email alerts and phone calls from the nurse care manager (NCM).
  Interventions: Behavioral: Nurse-led reminder program through email
- Management of diabetic patients (No Intervention): Usual care, educational program and usual management of Diabetic patients

INTERVENTIONS:
Behavioral: Nurse-led reminder program through email — Both groups will receive an educational program and usual care. The educational program will consist of:
  - 1-hour session, during which the NCM give advices and enphasize the importance of the correct procedure of glycemic control, report non-pharmacological strategies for a healty lifestyle and instruction on how to fill a self assessment form.
  Arms: Nurse-led email program through email

SUMMARY:
A number of strategies have been evaluated to improve clinical outcomes in diabetics patients, however no studies explored the efficacy of a nurse-led reminder program through email (NRP-e) to improve medication adherence, even if it is fundamental in the management of diabetics. The study aims at evaluating for the first time the efficacy of a nurse-led reminder program through email (NRP-e) to improve medication adherence in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

To be elegible, all subjects had to be diabetics (Diabetes Mellitus, Non-Insulin-Dependent)

* Speaking and reading italian
* Having an active phone number and an email address
* Providing a signed a informed consent

Exclusion Criteria:

* Mental illness
* Hospitalized patients and who refused to partecipate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 6 months
  The main outcome of the study was the improvement of medication adherence in diabetic patients between baseline and the end of follow-up.

SECONDARY OUTCOMES:
Trust in nurses | 6 months
  Mean differences between groups in the average scores of trust in nurses perceived by patients between baseline and the end of follow-up.
Lifestyle | 6 months
  Mean differences between groups in the average reduction in smoking and alcohol consumption, BMI and in the average increase of consumption of a healthy diet in diabetic patients between baseline and the end of follow-up.
Contacts with health services | 6 months
  Mean differences between groups in the reduction of the number of contact sand admissions of diabetic patients at health care services, between baseline and the end of follow-up.